CLINICAL TRIAL: NCT00964782
Title: The Effects of Sildenafil on Exercise Function and Capacity in Patients With Fontan Circulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 31171
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Fontan Circulation
Keywords: Fontan; sildenafil; exercise capacity; Patients with Fontan Circulation
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sildenafil crossover to placebo (Active Comparator): Sildenafil dosage (0.5mg/kg (max 20mg)) administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with treatment 2, placebo drug administered before the exercises.
  Interventions: Drug: Sildenafil; Drug: Placebo 2
- Placebo crossover to sidenafil (Placebo Comparator): Patient will receive a look-alike placebo administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with treatment 2 Sildenafil dosage will be 0.5mg/kg (max 20mg) administered before the exercises.
  Interventions: Drug: Placebo; Drug: Sildenafil 2

INTERVENTIONS:
Drug: Sildenafil — oral suspension, 0.5mg/kg, taken once prior to exercise stress test. Enrolled patients will be randomized to receive Sildenafil first and then crossed over to receive the opposite intervention, placebo.
  Other Names: Viagra
  Arms: Sildenafil crossover to placebo
Drug: Placebo — Patient will receive a look-alike placebo. Enrolled patients will be randomized to receive Placebo first and then crossed over to receive the opposite intervention, Sildenafil.
  Other Names: Ora-sweet and Ora-plus (1:1 ratio).
  Arms: Placebo crossover to sidenafil
Drug: Sildenafil 2 — oral suspension, 0.5mg/kg, taken once prior to exercise stress test. Enrolled patients will receive Sildenafil, the crossed over intervention from their initial intervention (Placebo).
  Other Names: Viagra
  Arms: Placebo crossover to sidenafil
Drug: Placebo 2 — Patient will receive a look-alike placebo. Enrolled patients will receive Placebo, the crossed over intervention from their initial intervention (Sildenafil).
  Other Names: Ora-sweet and Ora-plus (1:1 ratio).
  Arms: Sildenafil crossover to placebo

SUMMARY:
The study will test the hypothesis that a single dose of sildenafil can increase the exercise capacity of pediatric patients with a Fontan Circulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years
* Male or female
* Possess Fontan Circulation

Exclusion Criteria:

* Severe heart failure (New York Heart Ass. functional class IV)
* Evidence of Fontan pathway obstruction
* History of exercise-induced severe arrhythmias
* Pregnancy (known or suspected)
* Orthopedic limitations that prevent ambulation on a treadmill
* Use of nitroglycerin
* Herbal medications

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2012-05-24 (Actual); Study Completion 2012-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devyani Chowdhury, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject withdrew consent before being randomized and subsequent medication administered.
Groups:
- Sildenafil Crossover to Placebo: Sildenafil dosage (0.5mg/kg (max 20mg)) administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with the placebo drug administered before the exercises.
- Placebo Crossover to Sidenafil: Patient will receive a look-alike placebo administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with the Sildenafil dosage will be 0.5mg/kg (max 20mg) administered before the exercises.
Period: Overall Study
Arm/Group | Sildenafil Crossover to Placebo | Placebo Crossover to Sidenafil
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil Crossover to Placebo | Placebo Crossover to Sidenafil | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Change in Exercise Capacity Measured Via Maximum Oxygen Consumed During Exercise (VO2)
Description: A change in exercise capacity measured via maximum oxygen consumed during exercise (VO2). The measurement will be obtained from the Exercise Stress Test
Time Frame: baseline to 1 hour
Measure: Mean (Standard Error); unit: ml/min/kg
Arm/Group | Sildenafil Crossover to Placebo | Placebo Crossover to Sidenafil
Number analyzed (Participants) | 7 | 8
ml/min/kg
  Sildenafil VO2 | 39.4 (2.6) | 36.8 (2.4)
  Placebo VO2 | 41.2 (3.4) | 34.4 (2.8)

2. Primary Outcome: The Change in Exercise Capacity Measured Via Exercise Time
Description: A change in exercise capacity measured via exercise time (in minutes). The measurement will be obtained from the Exercise Stress Test
Time Frame: baseline to 1 hour
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Sildenafil Crossover to Placebo | Placebo Crossover to Sidenafil
Number analyzed (Participants) | 7 | 8
minutes
  Sildenafil Time | 11.6 (0.6) | 10.5 (0.4)
  Placebo Time | 12.1 (0.8) | 10.5 (0.5)

3. Secondary Outcome: The Change in Exercise Capacity Measured Via Maximum Heart Rate
Description: A change in exercise capacity measured via maximum heart rate (in beats per minute). The measurement will be obtained from the Exercise Stress Test
Time Frame: Baseline to 1 Hour
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Sildenafil Crossover to Placebo | Placebo Crossover to Sidenafil
Number analyzed (Participants) | 7 | 8
beats per minute
  Sildenafil Heart Rate | 182.3 (6.4) | 175.4 (6.9)
  Placebo Heart Rate | 182.6 (7.2) | 167.8 (7.0)

4. Secondary Outcome: The Change in Exercise Capacity Measured Via Minimum Oxygen Saturation Levels.
Description: A change in exercise capacity measured via minimum oxygen saturation (%). The measurement will be obtained from the Exercise Stress Test
Time Frame: Baseline to 1 Hour
Measure: Mean (Standard Error); unit: Percentage of oxygen saturation
Arm/Group | Sildenafil Crossover to Placebo | Placebo Crossover to Sidenafil
Number analyzed (Participants) | 7 | 8
Percentage of oxygen saturation
  Sildenafil minimum oxygen saturation % | 94.1 (1.0) | 94.6 (0.7)
  Placebo minimum oxygen saturation % | 93.1 (0.8) | 93.8 (0.6)

5. Secondary Outcome: The Change in Exercise Capacity Measured Via Metabolic Equivalents of Task (METs).
Description: A change in exercise capacity measured via metabolic equivalents of task (METs). The measurement will be obtained from the Exercise Stress Test. One MET is defined as 3.5 mL 02 uptake/kg per minute
Time Frame: Baseline to 1 hour
Measure: Mean (Standard Error); unit: Mets
Groups:
- Sildenafil: Sildenafil dosage (0.5mg/kg (max 20mg)) administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with the placebo drug administered before the exercises. This repeated test will occur on a separate date, not to exceed 3 months from baseline.
- Placebo: Patient will receive a look-alike placebo administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with the Sildenafil dosage will be 0.5mg/kg (max 20mg) administered before the exercises. This repeated test will occur on a separate date, not to exceed 3 months from baseline.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 7 | 8
Mets
  Sildenafil Metabolic Equivalent | 13.6 (0.7) | 12.4 (0.5)
  Placebo Metabolic Equivalent | 14.1 (0.9) | 12.1 (0.6)

ADVERSE EVENTS:
Groups:
- Sildenafil Crossed Over to Placebo: Sildenafil dosage (0.5mg/kg (max 20mg)) administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with the placebo drug administered before the exercises.
- Placebo Crossed Over to Sildenafil: Patient will receive a look-alike placebo administered at the time of enrollment followed by a battery of exercise tests. After a washout period, the process will be repeated with the Sildenafil dosage will be 0.5mg/kg (max 20mg) administered before the exercises.
Arm/Group | Sildenafil Crossed Over to Placebo | Placebo Crossed Over to Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil Crossed Over to Placebo (N=15) | Placebo Crossed Over to Sildenafil (N=15)
Flushed skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes